CLINICAL TRIAL: NCT02992288
Title: A Multicenter, Randomized, Placebo-controlled, Parallel Group, Double Blind, Dose-finding Phase II Trial to Study the Efficacy, Safety, Pharmacokinetic and Pharmacodynamic Effects of the Oral Partial Adenosine A1 Receptor Agonist Neladenoson Bialanate Over 20 Weeks in Patients With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: A Trial to Study Neladenoson Bialanate Over 20 Weeks in Patients With Chronic Heart Failure With Reduced Ejection Fraction
Acronym: PANTHEON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15128; 2016-003839-38 (EudraCT Number)
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
Keywords: Chronic Heart Failure; Heart Failure with Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — neladenoson bialanate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Neladenoson bialanate (BAY1067197) (5 mg) (Experimental): Chronic heart failure with reduced ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Neladenoson bialanate (BAY1067197) (10 mg) (Experimental): Chronic heart failure with reduced ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Neladenoson bialanate (BAY1067197) (20 mg) (Experimental): Chronic heart failure with reduced ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Neladenoson bialanate (BAY1067197) (30 mg) (Experimental): Chronic heart failure with reduced ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Neladenoson bialanate (BAY1067197) (40 mg) (Experimental): Chronic heart failure with reduced ejection fraction
  Interventions: Drug: Neladenoson bialanate (BAY1067197)
- Placebo (Placebo Comparator): Chronic heart failure with reduced ejection fraction
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neladenoson bialanate (BAY1067197) — 5 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (5 mg)
Drug: Neladenoson bialanate (BAY1067197) — 10 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (10 mg)
Drug: Neladenoson bialanate (BAY1067197) — 20 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (20 mg)
Drug: Neladenoson bialanate (BAY1067197) — 30 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (30 mg)
Drug: Neladenoson bialanate (BAY1067197) — 40 mg orally once daily for 20 weeks
  Arms: Neladenoson bialanate (BAY1067197) (40 mg)
Drug: Placebo — Orally once daily for 20 weeks
  Arms: Placebo

SUMMARY:
The objective of the study is to find the optimal dose of once daily oral neladenoson bialanate (BAY 1067197) when given in addition to standard therapy for heart failure with reduced ejection fraction (HFrEF).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and older
* Diagnosis of chronic heart failure (CHF), NYHA ( New York Heart Association ) class II-IV, LVEF ≤ 35% and elevated NT-proBNP

Exclusion Criteria:

* Acute de-novo heart failure
* Requirement of any intravenous (IV) treatments following 48 hours prior to randomization
* Mechanical support (e.g. intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device)
* Any cause of chronic heart failure other than ischemic cardiomyopathy and idiopathic dilated cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (75):
- United States (9):
  - Southwest Florida Research, Naples, Florida
  - Henry Ford Health System, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis Heart & Vascular, PC, St Louis, Missouri
  - Glacier View Research Institute-Cardiology, Kalispell, Montana
  - Stony Brook University Medical Center, Stony Brook, New York
  - St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - East Texas Cardiology, Houston, Texas
- Belgium (4):
  - AZ St-Jan Brugge Oostende AV, Bruges
  - Grand Hôpital de Charleroi, Gilly
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout
- Bulgaria (6):
  - Spec Hosp for Active Treatm in Cardiology Sv Georgi Pernik, Pernik
  - Specialized Hospital for Actrive Treatm of Card - Pleven, Pleven
  - NMTH Tzar Boris III, Sofia
  - UMHAT Tsaritsa Joanna-ISUL EAD Sofia, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Sofia, Sofia
  - MHAT Dr Stefan Cherkezov, Veliko Tarnovo
- Germany (6):
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Herz- und Diabeteszentrum Nordrhein-Westfalen (HDZ NRW), Bad Oeynhausen, North Rhine-Westphalia
  - St.-Johannes-Hospital Dortmund, Dortmund, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Charité Campus Virchow-Klinikum (CVK), Berlin
- Greece (5):
  - KAT General Hospital of Athens, Kifisia / Athens, Attica
  - G. Gennimatas General State Hospital of Athens, Athens
  - Thriassio General Hospital of Elefsina, Elefsina
  - Konstantopoulio General Hospital of Nea Ionia - Agia Olga, Nea Ionia / Athens
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
- Israel (7):
  - Barzilai Medical Center, Ashkelon
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Corporation, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Mount Scopus, Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Zrifin
- Italy (6):
  - A.O.U. Policlinico Federico II Napoli, Napoli, Campania
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - IRCCS Centro Cardiologico Fondazione Monzino, Milan, Lombardy
  - AUSL 8 Arezzo, Arezzo, Tuscany
- Japan (14):
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Takasaki General Medical C, Takasaki, Gunma
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - National hospital Organization Mito Medical Center, Higashiibaraki, Ibaraki
  - R.I.A.C Naha City Hospital, Naha, Okinawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Minamino Cardiovascular Hospital, Hachiōji, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Okayama Rosai Hospital, Okayama
  - Osaka General Medical Center, Osaka
  - Toyama Prefectural Central Hospital, Toyama
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Poland (7):
  - KLIMED Marek Klimkiewicz, Bialystok
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - Szpital Specjalistyczny im. J. Dietla, Krakow
  - Nzoz Salus, Lodz
  - Szpital Kliniczny Przemienienia Panskiego, Poznan
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - IV Wojskowy Szpital Kliniczny z Poliklinika, SPZOZ, Wroclaw
- Spain (7):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitario "Virgen de la Arrixaca", El Palmar, Murcia
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

REFERENCES:
- [Derived] Voors AA, Bax JJ, Hernandez AF, Wirtz AB, Pap AF, Ferreira AC, Senni M, van der Laan M, Butler J; PANTHEON Investigators. Safety and efficacy of the partial adenosine A1 receptor agonist neladenoson bialanate in patients with chronic heart failure with reduced ejection fraction: a phase IIb, randomized, double-blind, placebo-controlled trial. Eur J Heart Fail. 2019 Nov;21(11):1426-1433. doi: 10.1002/ejhf.1591. Epub 2019 Sep 16. PMID 31523892
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 11 countries between 22 February 2017 (first participant first visit) and 16 May 2018 (last participant last visit).
Pre-assignment Details: Overall, 462 participants were screened. Of them, 35 participants did not complete screening due to unmet eligibility criteria, consent withdrawal, adverse events and other unspecified reasons. In total, 427 participants were randomized and 426 participants received study treatment.
Groups:
- Placebo: Participants received placebo matched to neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 5 mg: Participants received 5 milligrams (mg) of neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 10 mg: Participants received 10 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 20 mg: Participants received 20 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 30 mg: Participants received 30 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 40 mg: Participants received 40 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
Period: Overall Study
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Started | 106 | 37 | 70 | 73 | 69 | 72
Treated | 106 | 37 | 70 | 72 | 69 | 72
Completed | 89 | 32 | 63 | 64 | 61 | 59
Not Completed | 17 | 5 | 7 | 9 | 8 | 13
Not completed — Adverse Event | 8 | 2 | 2 | 2 | 2 | 7
Not completed — Non-compliance with study drug | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 3 | 0 | 1 | 0 | 0 | 1
Not completed — Death | 2 | 0 | 2 | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg | Total
Number analyzed (Participants) | 106 | 37 | 70 | 73 | 69 | 72 | 427
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.9 (9.4) | 66.6 (10.5) | 66.4 (11.2) | 68.1 (10.0) | 67.6 (9.8) | 67.5 (10.0) | 67.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 11 | 14 | 12 | 7 | 71
  Male | 88 | 28 | 59 | 59 | 57 | 65 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 2 | 0 | 5
  Not Hispanic or Latino | 105 | 37 | 69 | 72 | 66 | 72 | 421
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 3 | 5 | 3 | 5 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 2 | 2 | 2 | 12
  White | 98 | 32 | 65 | 66 | 64 | 65 | 390
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: Percentage of LVEF] — Left ventricular ejection fraction (LVEF) is defined as the fraction of blood being pumped out of the left ventricle of the heart with each contraction.
  Percentage of LVEF | 28.24 (10.67) | 26.22 (7.99) | 27.58 (8.92) | 29.70 (10.87) | 29.87 (11.54) | 26.24 (8.92) | 28.18 (10.17)
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — NYHA classifies the extent of heart failure as Class I: Cardiac disease without resulting limitation of physical activity, Class II: Cardiac disease resulting in slight limitation of physical activity, Class III: Cardiac disease resulting in marked limitation of physical activity and Class IV: Cardiac disease resulting in inability to carry out any physical activity without discomfort.
  Participants
    Class I | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Class II | 62 | 23 | 38 | 44 | 49 | 49 | 265
    Class III/IV | 44 | 14 | 31 | 29 | 20 | 23 | 161
N-terminal pro-hormone b-type natriuretic peptide (NT-proBNP) [Median (Full Range); unit: Picograms per milliliter (pg/mL)] | 2111.00 [78.0 to 30428.0] | 2071.00 [155.0 to 17760.0] | 2063.00 [25.5 to 49896.0] | 1894.50 [56.0 to 13294.0] | 2084.00 [406.0 to 24551.0] | 2419.00 [60.0 to 13387.0] | 2085.00 [25.5 to 49896.0]
Medical history: Chronic heart failure etiology [Count of Participants; unit: Participants]
  Ischemic | 65 | 25 | 45 | 50 | 37 | 42 | 264
  Non-ischemic | 41 | 12 | 24 | 23 | 32 | 30 | 162
  Missing | 0 | 0 | 1 | 0 | 0 | 0 | 1
Medical history: Atrial fibrillation [Count of Participants; unit: Participants]
  With Atrial fibrillation | 44 | 14 | 27 | 26 | 27 | 33 | 171
  Without Atrial fibrillation | 62 | 23 | 43 | 47 | 42 | 39 | 256
Medication of interest: Beta-blocker [Count of Participants; unit: Participants]
  Beta-blocker | 103 | 37 | 66 | 70 | 67 | 69 | 412
  Not used at baseline | 3 | 0 | 4 | 3 | 2 | 3 | 15
Medication of interest: Angiotensin-converting enzyme inhibitor [Count of Participants; unit: Participants]
  Angiotensin-converting enzyme inhibitor | 58 | 19 | 41 | 41 | 36 | 45 | 240
  Not used at baseline | 48 | 18 | 29 | 32 | 33 | 27 | 187
Medication of interest: Angiotensin receptor blocker [Count of Participants; unit: Participants]
  Angiotensin receptor blocker | 15 | 6 | 11 | 14 | 9 | 9 | 64
  Not used at baseline | 91 | 31 | 59 | 59 | 60 | 63 | 363
Medication of interest: Angiotensin receptor-neprilysin inhibitor [Count of Participants; unit: Participants]
  Angiotensin receptor-neprilysin inhibitor | 20 | 7 | 9 | 9 | 12 | 12 | 69
  Not used at baseline | 86 | 30 | 61 | 64 | 57 | 60 | 358
Medication of interest: Mineralocorticoid receptor antagonist [Count of Participants; unit: Participants]
  Mineralocorticoid receptor antagonist | 93 | 33 | 56 | 60 | 56 | 57 | 355
  Not used at baseline | 13 | 4 | 14 | 13 | 13 | 15 | 72

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Left Ventricular Ejection Fraction (LVEF) (%) at Week 20 Measured by Echocardiography
Description: Left ventricular ejection fraction (LVEF) was measured by echocardiography. Mean and standard deviation were reported.
Time Frame: Baseline, Week 20
Population: Per-protocol set (PPS) included all participants without validity findings affecting efficacy evaluation. The participants with invalid/missing baseline or missing post-baseline LVEF values not due to cardiovascular (CV) death or heart failure (HF) hospitalization or with other major protocol deviation were excluded from PPS LVEF set.
Measure: Mean (Standard Deviation); unit: Percentage of LVEF
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 47 | 19 | 35 | 47 | 40 | 38
Percentage of LVEF | -2.19 (8.39) | 2.59 (8.48) | -3.01 (10.43) | 0.13 (8.74) | -2.45 (10.54) | 1.53 (10.01)
Statistical Analysis 1: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.2297, MCP-Mod method — Linear dose-response shape: The multiple comparison procedures (MCP) approach was applied to calculate the adjusted one-sided one-sided p-values of the contrast test; Dose response relationship was assessed using the MCP-Mod method combining MCP principles with modeling techniques under model uncertainty
Statistical Analysis 2: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.4409, MCP-Mod method — Sigmoidal Emax 1 dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.2842, MCP-Mod method — Sigmoidal Emax 2 dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.2534, MCP-Mod method — Emax dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.3842, MCP-Mod method — Quadratic dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Absolute Change From Baseline in Log-transformed NT-pro B-type Natriuretic Peptide (BNP) at Week 20
Description: NT-pro b-type Natriuretic Peptide (BNP) was measured. Mean and standard deviation were reported.
Time Frame: Baseline, Week 20
Population: PPS included all participants without validity findings affecting efficacy evaluation. The participants with invalid/missing baseline or missing post-baseline BNP value not due to CV death or HF hospitalization or with other major protocol deviation were excluded from the PPS BNP.
Measure: Mean (Standard Deviation); unit: log picograms per milliliter
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 82 | 29 | 58 | 59 | 53 | 56
log picograms per milliliter | -0.07 (0.70) | -0.24 (0.90) | -0.07 (0.52) | -0.07 (0.56) | 0.07 (0.55) | -0.08 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.8966, MCP-Mod method — Linear dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.9233, MCP-Mod method — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.9296, MCP-Mod method — [p-value comment as in outcome 1, analysis 3]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.7357, MCP-Mod method — [p-value comment as in outcome 1, analysis 4]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.9083, MCP-Mod method — [p-value comment as in outcome 1, analysis 5]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Left Ventricular End-Systolic Volume (LVESV) at Week 20
Description: LVESV was defined as the volume of blood in the left ventricle at the end of contraction, or systole and the beginning of filling or diastole. Mean and standard deviation were reported.
Time Frame: Baseline, Week 20
Population: PPS included all participants without validity findings affecting efficacy evaluation. The participants with invalid/missing baseline or missing post-baseline LVEF values not due to CV death or HF hospitalization or with other major protocol deviation were excluded from PPS LVEF set.
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 47 | 19 | 35 | 47 | 40 | 38
Milliliters (mL) | -5.44 (33.29) | -21.41 (48.13) | -2.82 (35.12) | -4.32 (29.73) | -3.12 (33.96) | -15.16 (39.65)
Statistical Analysis 1: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.4596, MCP-Mod method — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.7859, MCP-Mod method — Sigmoidal Emax1 dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.5562, MCP-Mod method — Sigmoidal Emax2 dose-response shape: The MCP approach was applied to calculate the adjusted one-sided p-values of the contrast test; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.5338, MCP-Mod method — [p-value comment as in outcome 1, analysis 4]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.7303, MCP-Mod method — [p-value comment as in outcome 1, analysis 5]; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Left Ventricular End-Diastolic Volume (LVEDV) at Week 20
Description: LVEDV was defined as the volume of blood in the left ventricle at end load or filling in diastole or the amount of blood in the ventricles just before systole. Mean and standard deviation were reported.
Time Frame: Baseline, Week 20
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliliters (mL)
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 47 | 19 | 35 | 47 | 40 | 38
Milliliters (mL) | -13.16 (40.23) | -21.65 (61.96) | -12.44 (39.84) | -5.92 (30.89) | -11.17 (42.32) | -19.69 (48.38)
Statistical Analysis 1: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.5703, MCP-Mod method — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.8253, MCP-Mod method — [p-value comment as in outcome 3, analysis 2]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.6506, MCP-Mod method — [p-value comment as in outcome 3, analysis 3]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.6923, MCP-Mod method — [p-value comment as in outcome 1, analysis 4]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.8036, MCP-Mod method — [p-value comment as in outcome 1, analysis 5]; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in High Sensitivity Troponin T (Hs-TNT) at Week 20
Description: High sensitivity troponin T (hs-TNT) was measured. Mean and standard deviation were reported.
Time Frame: Baseline, Week 20
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 82 | 29 | 58 | 59 | 53 | 56
Picograms per milliliter (pg/mL) | 0.13 (9.98) | 6.46 (33.04) | 3.77 (22.32) | 7.43 (37.79) | 2.59 (12.90) | 7.03 (24.81)
Statistical Analysis 1: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.9955, MCP-Mod method — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.9946, MCP-Mod method — [p-value comment as in outcome 3, analysis 2]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.9913, MCP-Mod method — [p-value comment as in outcome 3, analysis 3]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.9982, MCP-Mod method — [p-value comment as in outcome 1, analysis 4]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Neladenoson Bialanate 5 mg vs Neladenoson Bialanate 10 mg vs Neladenoson Bialanate 20 mg vs Neladenoson Bialanate 30 mg vs Neladenoson Bialanate 40 mg; Test type: Superiority; p = 0.9959, MCP-Mod method — [p-value comment as in outcome 1, analysis 5]; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Composite Efficacy Outcome
Description: Composite efficacy outcome was the first occurrence of CV death, HF hospitalization or urgent visit for HF. Number of participants with composite efficacy outcome were reported.
Time Frame: Baseline up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 82 | 29 | 58 | 59 | 53 | 56
Participants | 10 | 4 | 10 | 9 | 7 | 8

7. Secondary Outcome: Number of Participants With Cardiovascular (CV) Mortality
Description: Cardiovascular (CV) mortality was assessed. Number of participants with CV mortality were reported.
Time Frame: Baseline up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 82 | 29 | 58 | 59 | 53 | 56
Participants | 1 | 1 | 3 | 1 | 2 | 1

8. Secondary Outcome: Number of Participants With Heart Failure (HF) Hospitalization and Urgent Visits for Heart Failure (HF)
Description: Number of participants with HF hospitalization and urgent visits for HF were reported.
Time Frame: Baseline up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Neladenoson Bialanate 5 mg | Neladenoson Bialanate 10 mg | Neladenoson Bialanate 20 mg | Neladenoson Bialanate 30 mg | Neladenoson Bialanate 40 mg
Number analyzed (Participants) | 82 | 29 | 58 | 59 | 53 | 56
Participants | 10 | 4 | 9 | 8 | 5 | 8

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 26 weeks
Groups:
- Neladenoson Bialanate 5mg: Participants received 5 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 10mg: Participants received 10 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 20mg: Participants received 20 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 30mg: Participants received 30 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
- Neladenoson Bialanate 40mg: Participants received 40 mg of neladenoson bialanate tablets orally once daily for 20 weeks.
Arm/Group | Placebo | Neladenoson Bialanate 5mg | Neladenoson Bialanate 10mg | Neladenoson Bialanate 20mg | Neladenoson Bialanate 30mg | Neladenoson Bialanate 40mg
All-Cause Mortality (participants affected / at risk) | 8/106 | 1/37 | 5/70 | 1/72 | 2/69 | 2/72
Serious Adverse Events (participants affected / at risk) | 31/106 | 13/37 | 28/70 | 22/72 | 28/69 | 26/72
Other Adverse Events (participants affected / at risk) | 24/106 | 10/37 | 15/70 | 18/72 | 24/69 | 19/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=106) | Neladenoson Bialanate 5mg (N=37) | Neladenoson Bialanate 10mg (N=70) | Neladenoson Bialanate 20mg (N=72) | Neladenoson Bialanate 30mg (N=69) | Neladenoson Bialanate 40mg (N=72)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 15 (20) | 7 (8) | 12 (14) | 6 (10) | 10 (17) | 11 (16)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 5 (8) | 1 (1) | 2 (2) | 3 (7) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Oedema due to cardiac disease (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serratia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device function test (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial septal defect repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular assist device insertion (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implantable defibrillator replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device failure (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=106) | Neladenoson Bialanate 5mg (N=37) | Neladenoson Bialanate 10mg (N=70) | Neladenoson Bialanate 20mg (N=72) | Neladenoson Bialanate 30mg (N=69) | Neladenoson Bialanate 40mg (N=72)
Cardiac failure (Cardiac disorders) | 9 (9) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Asthenia (General disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 6 (8) | 1 (1)
Renal impairment (Renal and urinary disorders) | 6 (7) | 1 (1) | 0 (0) | 4 (4) | 6 (6) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (6) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 5 (6) | 4 (4) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 30 days but less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT02992288/SAP_000.pdf
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT02992288/Prot_001.pdf